CLINICAL TRIAL: NCT02643758
Title: Randomised Clinical Trial: Myopia Control Using Soft Bifocal Lenses
Brief Title: Myopia Control Using Soft Bifocal Lenses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A corporate decision to terminate the study
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Menicon Co., Ltd. (Industry); Queensland University of Technology (Other)
Responsible Party: Principal Investigator, Pauline Cho, Prof, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20151016008
Record Dates: First submitted 2015-12-08; First posted 2015-12-31 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Myopia
Keywords: Myopia control, bifocal soft contact lenses, children
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bifocal soft contact lenses (Experimental): Device: Bifocal soft contact lenses Use of bifocal contact lenses with nasally decentered optical zone to control the progression of myopia
  Interventions: Device: Bifocal soft contact lenses
- Single vision spectacles (No Intervention): Control: Single vision spectacles

INTERVENTIONS:
Device: Bifocal soft contact lenses
  Other Names: Menicon Duo 2 week soft bifocal lenses
  Arms: Bifocal soft contact lenses

SUMMARY:
The purpose of this study is to evaluate whether bifocal soft contact lenses (CLs) with low addition and nasally decentered optical zone are effective in controlling myopic progression in children. Visual manipulations induced by multifocal soft CLs with high addition have been shown to inhibit eye growth and myopia development in children by recent studies. Several theories have been proposed including alteration in peripheral defocus, reduced accommodation demand, alterations in binocular vision status and increased ocular higher order aberrations. However, those theories remain to be proven and the optical properties and performance of multifocal soft CLs have not been investigated in children.

DETAILED DESCRIPTION:
Visual manipulations induced by multifocal soft contact lenses (CLs) with high addition (+2.00 D or above) have been shown to inhibit eye growth and myopia development in children with up to 25-50% efficacy by recent studies. Several theories have been proposed including; alteration in peripheral defocus, reduced accommodation demand, alterations in binocular vision status and increased ocular higher order aberrations, which remain to be proven. However, the effect of controlling myopic progression by bifocal CLs with low addition has not been studied.

Several studies have shown that multifocal soft CLs can induce changes in ocular aberrations and degradation of image qualities in adults, whereas the optical properties and performance of multifocal soft CLs have not been investigated in children. Due to the differences in ocular structure and function, for instance, the pupil size and accommodation response, the performance of multifocal CLs in children may vary compared with that in adults. As a result, it is essential to assess the optical quality of these lenses worn by children for myopia control, through COAS (Complete Ophthalmic Analysis System).

The aim of this randomized clinical trial is to evaluate myopic progression in children wearing soft bifocal with low addition CLs (Menicon 2 week Duo **) used as daily disposable lenses, compared to control subjects wearing single-vision spectacles. Myopia progression quantified by changes in axial length (AL) and cycloplegic refractive error (Rx) will be monitored for 2 years with single-masking. The optical performance of bifocal CLs worn by children will also be investigated.

(**this lens is currently commercially available in Japan only. The oxygen permeability (Dk) is 34 with 72% water content, FDA group Ⅱ.)

ELIGIBILITY:
Inclusion Criteria:

* Refractive sphere: -0.75 D to -4.50 D
* Refractive cylinder: not exceed 1.00 D
* Spherical equivalent: -0.75 D to -5.00 D
* Best corrected distance VA (LogMAR): 0.14 or better in each eye and 0.10 or better in both eyes
* Difference in refractive error (spherical equivalent) in the two eyes: not exceed 1.00 D

Exclusion Criteria:

* Prior history of myopia control treatment
* Contraindication to contact lens wear
* Binocular anomalies (e.g. strabismus)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in axial length in 2 years | Every 6 months for a period of 2 years
  Evaluate the changes in cycloplegic axial length in children wearing bifocal soft contact lenses with low addition used as daily disposable lenses compared to control subjects wearing single-vision spectacles for two years with single masking and randomisation
Changes in cycloplegic refractive error in 2 years | Every 6 months for a period of 2 years
  Evaluate the changes in cycloplegic refractive error in children wearing bifocal soft contact lenses with low addition used as daily disposable lenses compared to control subjects wearing single-vision spectacles for two years with single masking and randomisation

SECONDARY OUTCOMES:
Changes in wavefront aberrations in 2 years | Every 6 months for a period of 2 years
  Assess changes in aberration profile by COAS (Complete Ophthalmic Analysis System) over a period of 2 years
Changes in accommodation responses in 2 years | Every 6 months for a period of 2 years
  Assess changes in the accommodation responses of children over a period of two years
Changes in wavefront aberrations of children with bifocal soft contact lenses in 2 years | Every 6 months for a period of 2 years
  Assess the aberration profile of children wearing bifocal soft contact lenses by COAS (Complete Ophthalmic Analysis System) over a period of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Cho, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Optometry, The Hong Kong Polytechnic University, Kowloon, Hong Kong

REFERENCES:
- [Background] Anstice NS, Phillips JR. Effect of dual-focus soft contact lens wear on axial myopia progression in children. Ophthalmology. 2011 Jun;118(6):1152-61. doi: 10.1016/j.ophtha.2010.10.035. Epub 2011 Jan 26. PMID 21276616
- [Background] Fujikado T, Ninomiya S, Kobayashi T, Suzaki A, Nakada M, Nishida K. Effect of low-addition soft contact lenses with decentered optical design on myopia progression in children: a pilot study. Clin Ophthalmol. 2014 Sep 23;8:1947-56. doi: 10.2147/OPTH.S66884. eCollection 2014. PMID 25284981
- [Background] Lam CS, Tang WC, Tse DY, Tang YY, To CH. Defocus Incorporated Soft Contact (DISC) lens slows myopia progression in Hong Kong Chinese schoolchildren: a 2-year randomised clinical trial. Br J Ophthalmol. 2014 Jan;98(1):40-5. doi: 10.1136/bjophthalmol-2013-303914. Epub 2013 Oct 29. PMID 24169657
- [Background] Sankaridurg P, Holden B, Smith E 3rd, Naduvilath T, Chen X, de la Jara PL, Martinez A, Kwan J, Ho A, Frick K, Ge J. Decrease in rate of myopia progression with a contact lens designed to reduce relative peripheral hyperopia: one-year results. Invest Ophthalmol Vis Sci. 2011 Dec 9;52(13):9362-7. doi: 10.1167/iovs.11-7260. PMID 22039230
- [Background] Walline JJ, Greiner KL, McVey ME, Jones-Jordan LA. Multifocal contact lens myopia control. Optom Vis Sci. 2013 Nov;90(11):1207-14. doi: 10.1097/OPX.0000000000000036. PMID 24061152
- [Background] Gifford P, Cannon T, Lee C, Lee D, Lee HF, Swarbrick HA. Ocular aberrations and visual function with multifocal versus single vision soft contact lenses. Cont Lens Anterior Eye. 2013 Apr;36(2):66-73; quiz 103-4. doi: 10.1016/j.clae.2012.10.078. Epub 2012 Nov 10. PMID 23146418
- [Background] Llorente-Guillemot A, Garcia-Lazaro S, Ferrer-Blasco T, Perez-Cambrodi RJ, Cervino A. Visual performance with simultaneous vision multifocal contact lenses. Clin Exp Optom. 2012 Jan;95(1):54-9. doi: 10.1111/j.1444-0938.2011.00666.x. Epub 2011 Nov 10. PMID 22070196